CLINICAL TRIAL: NCT04722731
Title: Prevention of Childhood Anxiety Disorders in Offspring of Anxious Parents - a Randomized Controlled Trial
Brief Title: Prevention of Childhood Anxiety Disorders in Offspring of Anxious Parents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Johan Åhlén, Project coordinator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JASE01
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Anxiety Disorders
Keywords: Prevention; Childhood anxiety; Parent program
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Confident Parents - Brave Children (Experimental): The Confident Parents - Brave Children (CPBT) is a group parent training targeted to anxious parents, delivered by a psychologist via video conference (the Zoom software solution).
  The CPBT will comprise six 120-minutes digital sessions. One month after the last group session, all parents will be offered to have an individual booster session with a psychologist over Zoom.
  Interventions: Behavioral: Confident Parents - Brave Children (CPBT)
- Self-help book (Active Comparator): In the control group, participants will receive a parenting book, titled "What all parents ought to know". This is a self-help book for parents, partly based on the scientifically evaluated parent program "All Children in Focus".
  Interventions: Behavioral: Self-help book "What all parents ought to know"

INTERVENTIONS:
Behavioral: Confident Parents - Brave Children (CPBT) — Session 1: Psychoeducation.
  Session 2: How to decrease criticism and rejection. Skills that provide a warm parenting style and acceptance of the child: validation and child directed play/activities.
  Session 3: Strategies to increase the autonomy of the child. The parents will learn how to use a stepladder approach to decrease overprotective behaviours.
  Session 4: How to decrease modelling of anxious behaviours and how to be a brave role model.
  Session 5: How to recognise and respond when your child is anxious. How to help your child approach new or scary things by using a stepladder approach.
  Session 6: Review of the principles and skills learned during the program. The group members will make a plan for how to continue the work on their own.
  Arms: Confident Parents - Brave Children
Behavioral: Self-help book "What all parents ought to know" — Participants in the control group will receive a self-help parenting book containing general research-based parenting strategies. They will be instructed to read the book within the 10 weeks from baseline to post.
  Arms: Self-help book

SUMMARY:
This study aims to expand the evidence of prevention of anxiety disorders in children. Children of anxious parents are at increased risk of developing anxiety disorders. Twin studies support a direct environmental transmission of anxiety between parent and child, and a main mechanism is suggested to be the parenting style of anxious parents, characterised by criticism and rejection, overprotection and modelling of anxiety.

This study will take a novel approach to prevent childhood anxiety disorders by evaluating the Confident Parents - Brave Children (CPBC) program, a parent program targeting anxious parents, in a randomised controlled trial (RCT).

DETAILED DESCRIPTION:
RESEARCH QUESTIONS

* Is the CPBC-program effective in preventing childhood anxiety disorders within a period of 12 and 36 months respectively, compared to a self-help parenting book?
* Is the CPBC-program effective in preventing childhood anxiety symptoms within a period of 12 and 36 months respectively, compared to a self-help parenting book?
* Is the effect moderated by severity of parental anxiety, child anxiety symptoms at baseline, or gender or age of the child?
* Is the study effective in increasing parental self efficacy?
* Is the effect of CPBC-program mediated by changes in parental criticism and rejection, overprotection, parental modelling of anxiety or parental accommodation?
* Is the CPBC-program cost-effective?

DESIGN The first study is a full scale parallel randomised controlled trial (allocation ratio 1:1). This study will include follow-up assessments after 12 and 36 months and will evaluate the relative efficacy of the CPBC-program versus an active control group (self-help book). The second part includes a mediation analysis and the third part is a within trial economic evaluation comparing the outcomes and costs between the CPBC-program and control using two types of analyses (cost-utility analysis and cost-consequence analysis).

POWER To have an 80% power to detect a significant (p ≤ 0.05) small to moderate difference (standardised mean difference = 0.4) the investigators will need to recruit 194 children. Given an anticipated attrition of 10%, the investigators will aim at including a total of 216 children. Participants will be recruited through advertisements. The participants will be randomly allocated to either (1) CPBC-program or (2) reading a self-help book.

ELIGIBILITY:
Inclusion Criteria:

1. The parent suffers from exaggerated worry or anxiety
2. The parent speaks and reads Swedish
3. The child is 5-9 years old
4. The child receives a clinicians assigned clinical severity rating (CSR) of 1 to 3 on anxiety disorders in ADIS-C (subclinical symptoms of anxiety)

Exclusion criteria:

1. Current or recent parental alcohol or substance abuse
2. The parent suffer from severe psychiatric conditions (e.g.current or recent psychotic or manic/hypomanic symptoms, severe depression or increased risk of suicide)
3. Social conditions that would obstruct from participation (e.g.ongoing custody dispute, domestic violence, ongoing investigation of child neglect through social services)
4. The child suffers from/is currently in treatment for an anxiety disorder or depression
5. The child is currently undergoing a neuropsychological evaluation
6. The child has no symptoms of anxiety at all (the child receives a clinicians assigned CSR of 0 on all anxiety disorders in the ADIS-C interview )
7. The child meet criteria for an anxiety disorder (the child receives a clinicians assigned CSR of 4 or above on any anxiety disorder in ADIS-C interview )

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 215 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in severity of childhood anxiety disorder as rated by clinician at 12-month, and 36 month follow-up | Base-line assessment, 12 month follow-up, 36 month follow-up
  Clinical Severity Ratings (CSR, ranging from 0 to 8, where a value of 4 and higher indicate that the child meet criteria for an anxiety disorder). The CSR is extracted from the Anxiety Disorders Interview Schedule - Schedule for Children (ADIS-C). The CRS is rated by clinician based on interviewing with primary caregiver.

SECONDARY OUTCOMES:
Change in Child Health Utility-9 Dimensions (CHU9D) at post-intervention, 12-month, and 36 month follow-up | Base-line assessment, post-intervention, 12 month follow-up, 36 month follow-up
  CHU9D is a validated parent-rated questionnaire of the child's quality of life, including 9 items (each item scored 1-5 where lower scores indicates better quality of life).
Change in EQ5D at post-intervention, at post-intervention, 12-month, and 36 month follow-up | Base-line assessment, post-intervention, 12 month follow-up, 36 month follow-up
  EQ5D is a validated self-rated questionnaire of the parent's quality of life, including 5 items (each item scored 1-3 where lower scores indicates better quality of life).
Change in Expressed Emotion Adjective Checklist (EEAC) at post-intervention, 12-month, and 36 month follow-up | Base-line assessment, post-intervention, 12 month follow-up, 36 month follow-up
  The EEAC is a validated self-rated questionnaire of the parent's positive and negative emotions directed towards the child. The EEAC include 20 adjectives (each scored 1-8 where 1 indicates never and 8 always.
Change in the Revised Parental Overprotective Scale (RPOS) at post-intervention, 12-month, and 36 month follow-up | Base-line assessment, post-intervention, 12 month follow-up, 36 month follow-up
  RPOS is a revised version of the validated self-rated questionnaire of the parent's overprotective behaviors, including 11 items (each item scored 1-5 where higher scores indicates more overprotective behaviors).
Change in the Modelling of Parental Anxiety Questionnaire (MPAQ) at post-intervention, 12-month, and 36 month follow-up | Base-line assessment, post-intervention, 12 month follow-up, 36 month follow-up
  MPAQ is a self-rated questionnaire of the parent's modelling of anxious and non-anxious behaviours (two different sub-scales), including 7+9 items (each item scored 1-5 where higher scores indicates more modelling).
Change in the Screen for Child Anxiety Related Disorders Revised (SCARED-R) at post-intervention, 12-month, and 36 month follow-up | Base-line assessment, post-intervention, 12 month follow-up, 36 month follow-up
  SCARED-R is a validated parent-rated questionnaire of the child's anxiety symptoms including 41 items (each item scored 0-2 where higher scores indicates more anxiety symptoms).
Change in the PHQ 9 at post-intervention, 12-month, and 36 month follow-up Change in the Patient Health Questionnaire (PHQ-9) at post-intervention, 12-month, and 36 month follow-up | Base-line assessment, post-intervention, 12 month follow-up, 36 month follow-up
  The PHQ-9 is a validated self-rated questionnaire of the parent's depression symptoms, including 9 items, (each item scored 0-3 where higher scores indicates more depressive symptoms).
Change in PROMIS-Anxiety Short Form at post-intervention, 12-month, and 36 month follow-up | Base-line assessment, post-intervention, 12 month follow-up, 36 month follow-up
  The PROMIS Anxiety Short Form is a validated self-rated questionnaire of the parent's anxiety symptoms, including 8 items, (each item scored 1-5 where higher scores indicates more anxiety symptoms).
Change in Family Accommodation Scale-Anxiety Parent Report (FASA-PR) at post-intervention, 12-month, and 36 month follow-up | Base-line assessment, post-intervention, 12 month follow-up, 36 month follow-up
  The FASA-PR is a validated self-rated questionnaire of the parent's accommodation to the child's anxiety, including 13 items (each item scored 0-4 where higher scores indicates more accommodation).
Change in Parenting Sense of Competence Scale (PSOC) at post-intervention, 12-month, and 36 month follow-up | Base-line assessment, post-intervention, 12 month follow-up, 36 month follow-up
  PSOC is a validated self-reported questionnaire of the parent's sense of competence, including 11 items (each item scored 1-6 where higher scores indicates more sense of competence).
Use of societal resources past three months (an adapted version of the TIC-P questionnaire) | Assessed at Base-line assessment, post-intervention, 12 month follow-up, 36 month follow-up
  TIC-P (Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness) is a questionnaire including questions about healthcare social support medications, parental absence from work, absence from school and productivity loss in school.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elfstrom S, Rosengren A, Andersson R, Engelbrektsson J, Isaksson A, Meregalli M, van Leuven L, Lalouni M, Ost LG, Ghaderi A, Ahlen J. Evaluating a program to prevent anxiety in children of anxious parents: a randomized controlled trial. J Child Psychol Psychiatry. 2025 Sep;66(9):1345-1356. doi: 10.1111/jcpp.14151. Epub 2025 Mar 12. PMID 40077809